CLINICAL TRIAL: NCT00017173
Title: Phase II Trial Of Surgery With Perioperative RPR/INGN 201 (Ad5CMV-p53) Gene Therapy Followed By Chemoradiotherapy For Advanced, Resectable Squamous Cell Carcinoma Of The Oral Cavity, Oropharynx, Larynx, and Pharynx
Brief Title: S0011, Gene Therapy & Surgery Followed by Chemo & RT in Newly Diagnosed Cancer of the Mouth or Throat
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068658; U10CA032102 (NIH); S0011 (Other: SWOG)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV verrucous carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — advexin; Cisplatin; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery with INGN 201 followed by chemo/RT (Experimental): intraoperative and postoperative injections of INGN 201 into the tumor bed, followed by cisplatin and radiation therapy
  Interventions: Biological: Ad5CMV-p53 gene; Drug: cisplatin; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: Ad5CMV-p53 gene — 2 intraoperative and one post-operative injection of Ad5CMV-p53.
  Other Names: INGN 201
Drug: cisplatin — 100 mg/m2 IV Day 1 every 21 days for 3 cycles
  Other Names: platinol
Procedure: conventional surgery — conventional surgery
  Other Names: surgery
Radiation: radiation therapy — 200 cGy per day Days 105 every week for 6 weeks
  Other Names: RT

SUMMARY:
RATIONALE: Inserting the p53 gene into a person's cancer cells may improve the body's ability to fight cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy with the p53 gene may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gene therapy plus surgery followed by cisplatin and radiation therapy in treating patients who have newly diagnosed resectable stage III or stage IV cancer of the mouth or throat.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of treating patients with newly diagnosed resectable stage III or IV squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx with surgery and Ad5CMV-p53 gene followed by cisplatin and radiotherapy.
* Determine the progression-free survival, local control, and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in this patient population.

OUTLINE: This is a multicenter study.

Patients undergo surgical resection and receive an intraoperative Ad5CMV-p53 gene injection into the resection bed and into the deep soft tissue bed of the cervical level with nodal metastasis. Patients also receive a third intraoperative Ad5CMV-p53 gene injection into the neck dissection bed, where it is allowed to sit in place for 10 minutes.

Within 48-72 hours after surgery, patients receive a postoperative Ad5CMV-p53 gene injection into each of two drainage catheters next to the mucosal suture line and neck dissection bed, where it is allowed to sit in place for 2 hours.

Within 56 days after surgery, patients receive cisplatin IV over 30-90 minutes on days 1, 22, and 43 and radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients may receive 3 additional days of radiotherapy to high-risk areas on days 43-45.

Patients are followed every 2-6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk/limited stage III or IV squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx

  * Newly diagnosed
  * Previously untreated
  * Considered surgically resectable
  * Evidence of regional lymph node metastases (N1-N3)
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 3 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine no greater than 2 times ULN
* Creatinine clearance at least 60 mL/min

Other:

* Magnesium normal (magnesium supplement allowed)
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* HIV negative
* Not pregnant or nursing
* Patients must use effective barrier contraception and prevent bodily fluid transmission during and for 28 days after Ad5CMV-p53 gene administration

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No concurrent intensity-modulated radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-02; Primary Completion 2007-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year
  accrual rate and percentage of patients successfully receiving the required doses of INGN 201

SECONDARY OUTCOMES:
Progression-free survival from time of registration until disease progression | two years
  percentage of patient who have not experience progression of disease at two years

CONTACTS AND LOCATIONS:
Overall Officials: George H. Yoo, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- [Derived] Yoo GH, Moon J, Leblanc M, Lonardo F, Urba S, Kim H, Hanna E, Tsue T, Valentino J, Ensley J, Wolf G. A phase 2 trial of surgery with perioperative INGN 201 (Ad5CMV-p53) gene therapy followed by chemoradiotherapy for advanced, resectable squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx: report of the Southwest Oncology Group. Arch Otolaryngol Head Neck Surg. 2009 Sep;135(9):869-74. doi: 10.1001/archoto.2009.122. PMID 19770418